CLINICAL TRIAL: NCT03533556
Title: Effects of L-theanine and Caffeine on Attention and Attention-related Brain Activity of Male Children and Adolescents With Attention Deficit Hyperactivity Disorder: a proof-of- Concept fMRI Study.
Brief Title: Effects of L-theanine and Caffeine on Attention and Attention-related Brain Activity of Children With Attention Deficit Hyperactivity Disorder
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Texas Tech University (Other)
Collaborators: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB2017-767
Record Dates: First submitted 2018-05-10; First posted 2018-05-23 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — theanine; Caffeine

STUDY DESIGN:
Intervention Model Description: 2.5 mg/kg body weight of L-theanine, 2.0 mg/kg body weight of caffeine and their combination each dissolved in 100 ml of water (solvent) or the solvent alone (i.e. placebo) will be administered on 4 separate days (at least 5 days apart) in a random counter-balanced order.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Dietary Supplement: L-theanine — Oral administration of 2.5 mg/kg body weight of L-theanine dissolved in 100 ml of water
Dietary Supplement: Caffeine — Oral administration of 2.0 mg/kg body weight of caffeine dissolved in 100 ml of water
Dietary Supplement: L-theanine-Caffeine Combination — Oral administration of a combination of 2.5 mg/kg body weight of L-theanine and 2.0 mg/kg body weight of caffeine dissolved in 100 ml of water
Other: Placebo — Oral administration of 100 ml of water

SUMMARY:
L-theanine and caffeine are two natural constituents of tea. Both of these compounds are among the U.S. Food and Drug Administration's list of Generally Recognized as Safe (GRAS) substances. Results of several clinical trials the PI and his team has conducted are consistent with results of many others to indicate that oral intake of each of 2.5 mg/kg body weight of L-theanine and 2.0 mg/kg body weight of caffeine is associated with improved attention in adults. Furthermore, there is evidence to suggest that, when taken in combination, L-theanine and caffeine seem to have additive effects in improving attention in adults. However, the specific actions of these substances have not been examined in children and adolescents with attention deficit hyperactivity disorder (ADHD), who are characterized by impaired attention, hyperkinesia and impulsivity.

Therefore, the investigators plan to study the functional activity of brains (both at rest and when performing standard tasks designed to measure attention) in children diagnosed with ADHD using functional magnetic resonance imaging, after they consume either 2.5 mg/kg of L-theanine, 2.0 mg/kg of caffeine and their combination as compared to a placebo (water). Based on our previous findings, the investigators expect to observe improvements (speed of responding and accuracy) in standard tests of attention with intake of L-theanine, caffeine and their combination as compared to the placebo. The investigators also expect to observe decreased functional activity in brain regions that typically show increased activity during mind wandering with intake of L-theanine, caffeine and their combination.

ELIGIBILITY:
Inclusion Criteria:

1. Children and adolescents (age 8-17 years)
2. Male
3. Diagnosed with ADHD by a clinician (e.g. a psychiatrist or a pediatrician)
4. Responded to stimulants (i.e. the symptoms of ADHD have improved in the past with a prescription of stimulants)

Exclusion Criteria:

1. Gross impairment of vision or hearing that would prevent the participants from performing neuropsychological tasks
2. Inability to read and follow written instructions
3. WISC-V IQ score of < 80
4. Physical, neurological or concurrent psychiatric impairments (except ADHD) that could affect cognitive and motor functions
5. Regular intake of medication that could alter visual, auditory, cognitive or motor functions (except stimulants)
6. History of head injury that resulted in loss of consciousness / history of brain surgery
7. Intake of drugs containing caffeine, other phosphodiesterase inhibitors or adenosine receptor blockers within the past 3 months
8. Intake of medications which are known to have pharmacological interactions with caffeine within the past 3 months
9. Current / past diagnosis of tics or other forms of dyskinesia
10. History of development of headache, drowsiness, anxiety, insomnia or nausea following intake of caffeine or caffeine containing beverages
11. Current / past history of smoking and / or alcohol or drug abuse
12. Absolute contraindications to undergo MRI
13. Unwillingness or inability to entirely refrain from use of electronic devices during study visits
14. Unwillingness or inability to refrain from intake of L-theanine and caffeine containing food or beverages within the 24 hours prior to each study visit
15. Unwillingness or inability to follow written, on-screen and verbal instructions given by the study team

Ages: 8 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity
Enrollment: 6 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Differences of fMRI blood oxygen level dependent (BOLD) responses of the brain in response to Stop Signals of an SSRT recorded following administration of each treatment and the placebo | 45 minutes after the administration of each treatment / placebo
  L-theanine, caffeine, L-theanine-caffeine combination and placebo will be administered on 4 separate days (at least 5 days apart) in a random counter-balanced order. Differences of functional magnetic resonance imaging reactivity of the whole brain, anterior and posterior nodes of the default mode network, bilateral dorsolateral prefrontal cortex and anterior cingulate cortex in response to stop signals of a stop signal reaction time task following administration of each treatment will be compared with the placebo.
Differences of fMRI blood oxygen level dependent (BOLD) responses of the brain in a Go-NoGo CPT recorded following administration of each treatment and the placebo | 60 minutes after the administration of each treatment / placebo
  L-theanine, caffeine, L-theanine-caffeine combination and placebo will be administered on 4 separate days (at least 5 days apart) in a random counter-balanced order. Differences of functional magnetic resonance imaging reactivity of the whole brain, anterior and posterior nodes of the default mode network, bilateral dorsolateral prefrontal cortex and anterior cingulate cortex in Go-NoGo continuous performance task following administration of each treatment will be compared with the placebo.
Differences of resting state fMRI functional connectivity recorded following administration of each treatment and the placebo | 75 minutes after the administration of each treatment / placebo
  L-theanine, caffeine, L-theanine-caffeine combination and placebo will be administered on 4 separate days (at least 5 days apart) in a random counter-balanced order. Differences of functional magnetic resonance imaging resting state functional connectivity of the anterior and posterior nodes of the default mode network, bilateral dorsolateral prefrontal cortex and anterior cingulate cortex and the remaining regions of the brain following administration of each treatment will be compared with the placebo.

SECONDARY OUTCOMES:
Differences of cerebral blood flow measured following administration of each treatment and the placebo | 80 minutes following administration of each treatment / placebo
  L-theanine, caffeine, L-theanine-caffeine combination and placebo will be administered on 4 separate days (at least 5 days apart) in a random counter-balanced order. Differences of cerebral blood flow estimated using arterial spin labeled echo following administration of each treatment will be compared with the placebo.
Differences of delay discounting following administration of each treatment and the placebo | 140 minutes following administration of each treatment / placebo
  L-theanine, caffeine, L-theanine-caffeine combination and placebo will be administered on 4 separate days (at least 5 days apart) in a random counter-balanced order. Differences of delay discounting as measured using a delay discounting task presented on a laptop computer following administration of each treatment will be compared with the placebo.
Differences of stop signal delay following administration of each treatment and the placebo | 45 minutes following administration of each treatment / placebo
  L-theanine, caffeine, L-theanine-caffeine combination and placebo will be administered on 4 separate days (at least 5 days apart) in a random counter-balanced order. Differences of stop signal delay of a stop signal reaction time task performed in the magnetic resonance imaging scanner following administration of each treatment will be compared with the placebo.
Differences of reaction times of correct Go responses in a Go-NoGo CPT following administration of each treatment and the placebo | 60 minutes following administration of each treatment / placebo
  L-theanine, caffeine, L-theanine-caffeine combination and placebo will be administered on 4 separate days (at least 5 days apart) in a random counter-balanced order. Differences of reaction times of correct Go responses in a Go-NoGo continuous performance task performed in the magnetic resonance imaging scanner following administration of each treatment will be compared with the placebo.
Differences of commission errors in the Go-NoGo CPT following administration of each treatment and the placebo | 60 minutes following administration of each treatment / placebo
  L-theanine, caffeine, L-theanine-caffeine combination and placebo will be administered on 4 separate days (at least 5 days apart) in a random counter-balanced order. Differences of commission errors in the Go-NoGo continuous performance task performed in the magnetic resonance imaging scanner following administration of each treatment will be compared with the placebo.
Differences of performance in Flanker Inhibitory Control and Attention Test following administration of each treatment and the placebo | 100 minutes following administration of each treatment / placebo
  L-theanine, caffeine, L-theanine-caffeine combination and placebo will be administered on 4 separate days (at least 5 days apart) in a random counter-balanced order. Differences of performance in Flanker Inhibitory Control and Attention Test of the NIH Toolbox Cognition Battery following administration of each treatment will be compared with the placebo.
Differences of performance in Dimensional Change Card Sort Test following administration of each treatment and the placebo | 100 minutes following administration of each treatment / placebo
  L-theanine, caffeine, L-theanine-caffeine combination and placebo will be administered on 4 separate days (at least 5 days apart) in a random counter-balanced order. Differences of performance in Dimensional Change Card Sort Test of the NIH Toolbox Cognition Battery following administration of each treatment will be compared with the placebo.
Differences of performance in Pattern Comparison Processing Speed Test following administration of each treatment and the placebo | 100 minutes following administration of each treatment / placebo
  L-theanine, caffeine, L-theanine-caffeine combination and placebo will be administered on 4 separate days (at least 5 days apart) in a random counter-balanced order. Differences of performance in Pattern Comparison Processing Speed Test of the NIH Toolbox Cognition Battery following administration of each treatment will be compared with the placebo.
Differences of post- vs. pre-treatment change of STAI-CH State Scale following administration of each treatment and the placebo | Immediately before and 90 minutes after administration of each treatment / placebo
  L-theanine, caffeine, L-theanine-caffeine combination and placebo will be administered on 4 separate days (at least 5 days apart) in a random counter-balanced order. Differences of State Trait Anxiety Inventory for Children (State Questionnaire) immediately prior to and following administration of each treatment will be compared with the corresponding post- vs. pre-treatment change of placebo.

OTHER OUTCOMES:
Differences of commission errors in SSRT following administration of each treatment and the placebo | 45 minutes following administration of each treatment / placebo
  L-theanine, caffeine, L-theanine-caffeine combination and placebo will be administered on 4 separate days (at least 5 days apart) in a random counter-balanced order. Differences of commission errors of the stop signal reaction time task performed in the magnetic resonance imaging scanner following administration of each treatment will be compared with the placebo.
Differences of omission errors in SSRT following administration of each treatment and the placebo | 45 minutes following administration of each treatment / placebo
  L-theanine, caffeine, L-theanine-caffeine combination and placebo will be administered on 4 separate days (at least 5 days apart) in a random counter-balanced order. Differences of omission errors of the stop signal reaction time task performed in the magnetic resonance imaging scanner following administration of each treatment will be compared with the placebo.
Differences of omission errors in Go-NoGo CPT following administration of each treatment and the placebo | 60 minutes following administration of each treatment / placebo
  L-theanine, caffeine, L-theanine-caffeine combination and placebo will be administered on 4 separate days (at least 5 days apart) in a random counter-balanced order. Differences of omission errors of the Go-NoGo continuous performance task performed in the magnetic resonance imaging scanner following administration of each treatment will be compared with the placebo.
Differences of performance in Picture Sequence Memory Test following administration of each treatment and the placebo | 100 minutes following administration of each treatment / placebo
  L-theanine, caffeine, L-theanine-caffeine combination and placebo will be administered on 4 separate days (at least 5 days apart) in a random counter-balanced order. Differences of performance in Picture Sequence Memory Test of the NIH Toolbox Cognition Battery following administration of each treatment will be compared with the placebo.
Differences of performance in List Sorting Working Memory Test following administration of each treatment and the placebo | 100 minutes following administration of each treatment / placebo
  L-theanine, caffeine, L-theanine-caffeine combination and placebo will be administered on 4 separate days (at least 5 days apart) in a random counter-balanced order. Differences of performance in List Sorting Working Memory Test of the NIH Toolbox Cognition Battery following administration of each treatment will be compared with the placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Chanaka Kahathuduwa, MBBS PhD, Principal Investigator — Texas Tech University
Locations (1):
- Texas Tech University - Department of Human Development and Family Studies, Lubbock, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided